CLINICAL TRIAL: NCT03101527
Title: Open Trial Determining Antidepressant Effects of Omega-3 Supplementation During Pregnancy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: William Coryell (Other)
Responsible Party: Sponsor-Investigator, William Coryell, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201002781
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder in Pregnancy
Keywords: Major Depressive Disorder; omega-3 polyunsaturated fatty acid; PUFA; Pregnancy; eicosapentaenoic acid (EPA) supplementation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: A single group model was used: pregnant women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supplementation (Experimental): Subjects received Omega-3 PUFA supplementation
  Interventions: Drug: Omega-3 PUFA supplementation

INTERVENTIONS:
Drug: Omega-3 PUFA supplementation — Subjects received 2.2g of eicosapentaenoic acid (EPA) and 1.2g docosahexaenoic daily for the duration of the study
  Other Names: eicosapentaenoic acid (EPA); docosahexaenoic acid (DHA)

SUMMARY:
The purpose of this study is to determine if omega-3 polyunsaturated fatty acids as a monotherapy have antidepressant effects during pregnancy. It will also provide pilot data pertaining to relationships between apparent response to omega-3 monotherapy and both plasma cytokine and erythrocyte essential fatty acid concentrations.

DETAILED DESCRIPTION:
Pregnancy does not reduce the risk of recurrence among women who have previously experienced depressive illness and the advent of new episodes during pregnancy raises particular problems. Lingering concerns over the possible teratogenicity of medications in general leave many women reluctant to continue preexisting antidepressant prophylaxis or to accept new trials of conventional antidepressant treatment. There is also now accumulating evidence that the SSRIs have short-, and perhaps longer-term, adverse effects on the newborn.

The antidepressant effects of omega-3 polyunsaturated fatty acid (PUFA) supplementation may offer a particularly appropriate alternative to conventional therapy for depressive episodes that occur during pregnancy. The nutritional needs of the fetus increase the likelihood of omega-3 PUFA deficits in the mother but access to adequate omega-3 PUFAs through fish intake is limited due to concerns over mercury levels. Because polyunsaturated fatty acids are dietary components essential for both fetal development and maternal health, and because their use as supplementation carries a minimal to non-existent side effect burden, women may be more likely to accept omega-3 supplementation over that of conventional antidepressants to manage depressive illness if provided sufficient evidence for effectiveness.

Data supporting the antidepressant potential of omega-3 PUFA supplementation derive first from numerous case-control studies that have associated depressive illness with lower tissue concentrations of omega-3 PUFAs and with higher ratios of omega-6 to omega-3. These findings prompted antidepressant trials of omega-3 supplementation as augmentation or as mono-therapy and many reports described significant benefits over placebo, including one that targeted pregnant women and yielded a large effect size. A number of other trials, however, failed to show clear antidepressant effects. Meta-analyses have highlighted these inconsistencies in results but have found no explanations for them in differing sample demographics, baseline depressive severity levels, PUFA dosing, or trial durations. Other sources of study outcome differences undoubtedly exist and a clear possibility is that the studies with positive results involved subjects more likely to truly benefit from omega-3 supplementation. The characteristics of such individuals are entirely unknown. Though valid predictors of antidepressant response to omega-3 PUFA supplementation would provide powerful tools for personalizing treatment no study has sought to identify them.

One feature that might characterize an individual likely to respond to omega-3 PUFA supplementation is, of course, the presence of relatively low tissue concentrations of omega-3 PUFAs and/or high ratios of omega-6 to omega-3 concentrations. The likelihood that omega-3 PUFA supplementation exerts antidepressant effects via modulation of the inflammatory cascade, and the extensive evidence that high levels of pro-inflammatory markers characterize individuals with depressive disorders, indicate that these measures too may help to select those most likely to benefit from treatment with omega-3 PUFAs.

The identification of response predictors for a specific antidepressant strategy would not only have value for the selection of acute treatment for individuals with active depression but could also be used to choose preventative strategies for individuals who are not currently depressed but who are at high risk because of a recent history of a depressive episode. Prophylaxis against depressive illness in such individuals would have special importance during pregnancy. The adverse effects of depressive illness on both maternal and newborn well-being are widely appreciated but women who develop depressive disorders during pregnancy may, for a variety of reasons, fail to report symptoms to their health care provider or, if they do, treatment response may be delayed or even absent after one or more trials.

ELIGIBILITY:
Inclusion Criteria:

1. Women with uncomplicated pregnancy within the 1st or 2nd trimester of pregnancy
2. Score of 10 or greater on the nine item Patient Health Questionnaire (PHQ-9) for depression

Exclusion Criteria:

1. antidepressant use in preceding month
2. use in previous 4 weeks of psychotropic medications other than hypnotics or benzodiazepines in diazepam dose-equivalents greater than or equal to 2mg/day for insomnia
3. Fish allergy
4. initiation of regularly scheduled course of psychotherapy within previous 2 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is focused on pregnant women.
Enrollment: 3 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The Hamilton Rating Scale for Depression (HAM-D) | Subjects were administered the HAM-D at Day 1 and every month thereafter until week 38 of their pregnancies.
  The HAM-D is a multiple item semi-structured clinician administered questionnaire used to assess the range, type and severity of depressive symptoms observed in patients with MDD. The HAM-D24 consists of 24 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-24 total score is calculated as the sum of the 24 individual symptom scores; the total score can range from 0 to 76. Higher HAMD-24 scores indicate more severe depression.
Montgomery-Asberg Depression Scale (MADRS) | Subjects were administered the MADRS on Day 1 and every month thereafter until week 38 of their pregnancies.
  The MADRS is a clinician administered semi-structured scaled designed to detect changes in depressive symptoms. The scale contains 10 items and ratings are graded from 0 to 6 , with 0 representing an absence of a symptom and 6 corresponding to the most severe degree of MDD symptomology.
Edinburgh Postnatal Depression Scale (EPDS) | Subjects were asked to complete the EPDS on Day 1 and every month thereafter until week 38 of their pregnancies
  The EPDS is a self-administered depression screen for postpartum women. The EPDS consists of 10 questions. Responses are scored 0,, 1, 2, or 3 according to increased severity of the symptom. Items marked with an * are reversed scored. A total score of 13 or more suggests follow-up intervention is warranted.
Beck Depression Scale (BDI) | Subjects were asked to complete the BDI on Day 1 and every month thereafter through week 38 of their pregnancies
  The BDI is a self-administered questionnaire developed to detect, assess, and monitor changes in depressive symptoms. It is composed of 21 items, each with 4 possible responses scored from 0 to 3 with 3 indicating a higher level of severity. For people who have been clinically diagnosed, scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression.

IPD SHARING:
Plan to Share IPD: No
The Investigator does not intend to share IPD

REFERENCES:
- [Background] Hibbeln JR. Seafood consumption, the DHA content of mothers' milk and prevalence rates of postpartum depression: a cross-national, ecological analysis. J Affect Disord. 2002 May;69(1-3):15-29. doi: 10.1016/s0165-0327(01)00374-3. PMID 12103448
- [Background] De Vriese SR, Christophe AB, Maes M. Lowered serum n-3 polyunsaturated fatty acid (PUFA) levels predict the occurrence of postpartum depression: further evidence that lowered n-PUFAs are related to major depression. Life Sci. 2003 Nov 7;73(25):3181-7. doi: 10.1016/j.lfs.2003.02.001. PMID 14561523
- [Background] Peet M, Murphy B, Shay J, Horrobin D. Depletion of omega-3 fatty acid levels in red blood cell membranes of depressive patients. Biol Psychiatry. 1998 Mar 1;43(5):315-9. doi: 10.1016/s0006-3223(97)00206-0. PMID 9513745
- [Background] Rees AM, Austin MP, Owen C, Parker G. Omega-3 deficiency associated with perinatal depression: case control study. Psychiatry Res. 2009 Apr 30;166(2-3):254-9. doi: 10.1016/j.psychres.2007.12.011. Epub 2009 Mar 5. PMID 19268372